CLINICAL TRIAL: NCT05761509
Title: "Observational Study on Tolerability and Observance of Post-exposure Prophylaxis With Doravirine in HIV Viral Risk"
Acronym: DORASPEP
Status: Completed | Type: Observational
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IMEA 067; N° IDRCB: 2022-A02325-38 (Other: ANSM, France)
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
Keywords: HIV; PEP; Doravirine; HIV exposure; HIV prevention
MeSH Terms: conditions — HIV Infections | interventions — doravirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: 200 subjects exposed to HIV, leading to prescription of 28-day doravirine based post exposure prophylaxis (PEP).
  The study referred to treatments that are using routinely in the medical care of subjects under PEP. These treatments are the following:
  * Delstrigo®: Fixed-dose combination containing 100mg of doravirine, 245 mg of tenofovir disoproxil and 300 mg of lamivudine, one tablet to be taken orally once daily, with or without food.
  * Pifeltro®: doravirine dosed at 100 mg, on tablet to be taken orally once daily, with or without food, in combination with tenofovir disoproxil/emtricitabine.
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — The study treatments will used during 28 days according to the routine care of each investigator center.
  Other Names: Delstrigo®; Pifeltro®

SUMMARY:
The main objective of this observational study is to assess the adherence of post exposure prophylaxis treatment with doravirine (using Delstrigo® or Pifeltro®), prescribed to subjects exposed to HIV according to French national recommendations.

This study will evaluate:

* the percentage of subjects who followed their treatment within the prescribed 28 days,
* the prevalence and type of side effects in subjects on this treatment,
* the occurrence of HIV seroconversion associated with this combination.

DETAILED DESCRIPTION:
The study visits are those routinely performed in the standard care of the subjects using PEP and are the following:

Visit 1 (between day 1 to day 8 after PEP treatment initiation):

* Subject information and inclusion in the study,
* Pregnancy test (urine or serum) for women of childbearing potential (WOCBP)
* Delivery of a follow-up subject diary (daily information about PEP treatment intake, concomitant treatments and potential side effects/adverse events)

Visit 2 (From 42 days to 90 days after PEP treatment initiation)

* Treatment observance (PEP),
* Return of the follow-up subject diary,
* Check of the follow-up subject diary completion,
* Keep a copy of the HIV serology and/or viral load results in the medical file.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years old
2. Exposure to HIV, leading to the prescription of 28-day post exposure prophylaxis (PEP)
3. PEP with doravirine:

   1. Delstrigo® (tenofovir disoproxil, doravirine, lamivudine),
   2. Or Pifeltro® (doravirine) in association with tenofovir disoproxil/emtricitabine.
4. Participant who can understand, read and speak French.
5. With or without health insurance.
6. Cisgender female and Female to Male transgender participants are eligible to participate if they are not pregnant or breastfeeding, and at least one of the following conditions applies: •

   1. Is not a WOCBP (Women Of Childbearing Potential) OR
   2. Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), or be abstinent as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the treatment period and for at least 8 weeks after the last dose. The investigator should evaluate the potential for contraceptive method failure (i.e., non compliance, recently initiated) in relationship to the first dose of PEP treatment.

A WOCBP must have a negative pregnancy test (urine or serum) before inclusion in the study. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant should not be included in the study if the serum pregnancy result is positive.

Exclusion Criteria:

1. Contraindication to Delstrigo® or Pifeltro® or tenofovir disoproxil/emtricitabine: hypersensitivity to active substances or excipients.
2. Contra-indicated treatment likely to interfere with the study drugs as listed in the summary of the product characteristics.
3. Viral resistance of the source subject known and unsuitable for the prescription of doravirine
4. Simultaneous participation in another clinical trial with an experimental treatment or any intervention, which may have impact/change onto the PEP treatments or within an exclusion period of a previous clinical trial at screening.
5. Subjects under legal guardianship or unable to express their consent.
6. Subject privated of liberty by judicial or administrative decision or subject under psychiatric care or admitted to a health or social establishment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects exposed to HIV, leading to the prescription of 28-day post exposure prophylaxis (PEP) with doravirine.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
To assess the adherence of post exposure prophylaxis treatment with doravirine (using Delstrigo® or Pifeltro®), prescribed to subjects exposed to HIV according to French national recommendations. | 3 months
  Proportion of subjects who complete the total period of treatment (intake during 28 days).
  The treatment completeness will be defined as follows:
  * no missing treatment intake from D1 to D14,
  * and no more than 2 missing treatment intakes from D15 to D28.

SECONDARY OUTCOMES:
To evaluate the tolerability of PEP with doravirine. | 28 days
  Number and type of side effects.
To evaluate the prevalence of HIV seroconversion associated with this combination. | 3 months
  Number of subjects with seroconversion.
To compare the adherence of post exposure prophylaxis treatment between Delstrigo® or Pifeltro® | 28 days
  Proportion of subjects who complete the total period of each treatment (intake during 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Karine Lacombe, Pr, Principal Investigator — Infectious diseases unit / Saint Antoine hospital, Paris (France); Roland Tubiana, MD, Principal Investigator — Infectious diseases unit / La Pitié-Salpêtrière hospital, Paris (France); Alain Makinson, Pr, Principal Investigator — Infectious diseases unit / Montpellier hospital, Montpellier (France)
Locations (3):
- France (3):
  - Service de maladies infectieuses et tropicales du CHU de Montpellier, Montpellier
  - Hopital Saint Antoine, Paris
  - Service de maladies infectieuses et tropicales de de l'hôpital La Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No
Will be decided later by the scientific committee.

REFERENCES:
- [Background] Rapport Morlat : Prise en charge des accidents d'exposition sexuelle et au sang (AES) chez l'adulte et l'enfant (septembre 2017) https://cns.sante.fr/wp-content/uploads/2017/10/experts-vih_aes.pdf.
- [Background] Assoumou L, Bocket L, Pallier C, Grude M, Ait-Namane R, Izopet J, Raymond S, Charpentier C, Visseaux B, Wirden M, Trabaud MA, Le Guillou-Guillemette H, Allaoui C, Henquell C, Krivine A, Dos Santos G, Delamare C, Bouvier-Alias M, Montes B, Ferre V, De Monte A, Signori-Schmuck A, Maillard A, Morand-Joubert L, Tumiotto C, Fafi-Kremer S, Amiel C, Barin F, Marque-Juillet S, Courdavault L, Vallet S, Beby-Defaux A, de Rougemont A, Fenaux H, Avettand-Fenoel V, Allardet-Servent A, Plantier JC, Peytavin G, Calvez V, Chaix ML, Descamps D; ANRS AC-43 Resistance Study Group. Stable prevalence of transmitted drug resistance mutations and increased circulation of non-B subtypes in antiretroviral-naive chronically HIV-infected patients in 2015/2016 in France. J Antimicrob Chemother. 2019 May 1;74(5):1417-1424. doi: 10.1093/jac/dkz011. PMID 30753724
- [Background] Pham HT, Xiao MA, Principe MA, Wong A, Mesplede T. Pharmaceutical, clinical, and resistance information on doravirine, a novel non-nucleoside reverse transcriptase inhibitor for the treatment of HIV-1 infection. Drugs Context. 2020 Mar 3;9:2019-11-4. doi: 10.7573/dic.2019-11-4. eCollection 2020. PMID 32180823
- [Background] Valin N, Fonquernie L, Daguenel A, Campa P, Anthony T, Guiguet M, Girard PM, Meyohas MC. Evaluation of tolerability with the co-formulation elvitegravir, cobicistat, emtricitabine, and tenofovir disoproxil fumarate for post-HIV exposure prophylaxis. BMC Infect Dis. 2016 Nov 29;16(1):718. doi: 10.1186/s12879-016-2056-3. PMID 27894270
- [Background] Inciarte A, Leal L, Gonzalez E, Leon A, Lucero C, Mallolas J, Torres B, Laguno M, Rojas J, Martinez-Rebollar M, Gonzalez-Cordon A, Cruceta A, Arnaiz JA, Gatell JM, Garcia F; STRIBPEP Study Group. Tenofovir disoproxil fumarate/emtricitabine plus ritonavir-boosted lopinavir or cobicistat-boosted elvitegravir as a single-tablet regimen for HIV post-exposure prophylaxis. J Antimicrob Chemother. 2017 Oct 1;72(10):2857-2861. doi: 10.1093/jac/dkx246. PMID 29091217
- [Background] Gantner P, Hessamfar M, Souala MF, Valin N, Simon A, Ajana F, Bouvet E, Rouveix E, Cotte L, Bani-Sadr F, Hustache-Mathieu L, Lebrette MG, Truchetet F, Galempoix JM, Piroth L, Pellissier G, Muret P, Rey D; E/C/F/TAF PEP Study Group. Elvitegravir-Cobicistat-Emtricitabine-Tenofovir Alafenamide Single-tablet Regimen for Human Immunodeficiency Virus Postexposure Prophylaxis. Clin Infect Dis. 2020 Feb 14;70(5):943-946. doi: 10.1093/cid/ciz577. PMID 31804669
- [Background] Eviplera: Product information from the European Medecines Agency: https://www.ema.europa.eu/en/medicines/human/EPAR/eviplera
- [Background] Genvoya: Product information from the European Medecines Agency: https://www.ema.europa.eu/en/medicines/human/EPAR/genvoya
- [Background] Pifeltro: Product information from the European Medecines Agency: https://www.ema.europa.eu/en/medicines/human/EPAR/pifeltro
- [Background] Delstrigo: Product information from the European Medecines Agency: https://www.ema.europa.eu/en/medicines/human/EPAR/delstrigo#product-information-section
- [Background] HIV drugs interactions, University of Liverpool: http://www.hiv-druginteractions.org
- [Background] Scheibe K, Urbanska A, Jakubowski P, Hlebowicz M, Bociaga-Jasik M, Raczynska A, Szymczak A, Szetela B, Lojewski W, Parczewski M. Low prevalence of doravirine-associated resistance mutations among polish human immunodeficiency-1 (HIV-1)-infected patients. Antivir Ther. 2021 May;26(3-5):69-78. doi: 10.1177/13596535211043044. Epub 2021 Oct 20. PMID 35485331
- [Background] Asante-Appiah E, Lai J, Wan H, Yang D, Martin EA, Sklar P, Hazuda D, Petropoulos CJ, Walworth C, Grobler JA. Impact of HIV-1 Resistance-Associated Mutations on Susceptibility to Doravirine: Analysis of Real-World Clinical Isolates. Antimicrob Agents Chemother. 2021 Nov 17;65(12):e0121621. doi: 10.1128/AAC.01216-21. Epub 2021 Sep 27. PMID 34570651
- See also: Eviplera: Product information from the European Medecines Agency — https://www.ema.europa.eu/en/medicines/human/EPAR/eviplera
- See also: Genvoya: Product information from the European Medecines Agency — https://www.ema.europa.eu/en/medicines/human/EPAR/genvoya
- See also: Pifeltro: Product information from the European Medecines Agency — https://www.ema.europa.eu/en/medicines/human/EPAR/pifeltro
- See also: Delstrigo: Product information from the European Medecines Agency — https://www.ema.europa.eu/en/medicines/human/EPAR/delstrigo
- See also: HIV drugs interactions, University of Liverpool — https://www.hiv-druginteractions.org/